CLINICAL TRIAL: NCT00929747
Title: Comparison of Corneal Aberrations and Visual Outcomes in AcrySof IQ Toric Patients Versus LRI Patients
Brief Title: Comparison of Corneal Aberrations and Visual Outcomes in AcrySof IQ Toric Patients Versus Limbal Relaxing Incision (LRI) Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M08-008
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2009-10

CONDITIONS: Cataracts
Keywords: Cataract; Toric; IOL; AcrySof, LRI
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toric IOL (Active Comparator): AcrySof IQ Toric IOL
  Interventions: Device: Toric
- Limbal Relaxing Incision (Active Comparator): AcrySof IQ with Limbal Relaxing Incision
  Interventions: Procedure: Limbal Relaxing Incision

INTERVENTIONS:
Device: Toric — Unilateral implantation of the AcrySof IQ Toric IOL
  Arms: Toric IOL
Procedure: Limbal Relaxing Incision — Unilateral implantation of a AcrySof IQ (SN60WF) IOL with concomitant LRI at the time of surgery
  Arms: Limbal Relaxing Incision

SUMMARY:
A prospective evaluation of postoperative corneal aberrations and visual parameters in patients assigned to either an AcrySof IQ Toric intraocular lens (IOL) group or a group implanted with a SN60WF IOL and having concomitant limbal relaxing incision.

ELIGIBILITY:
Inclusion Criteria:

1. operable cataracts
2. good ocular health
3. 0.5 D to 2.0 D of corneal astigmatism

Exclusion Criteria:

1. > 2.0 D astigmatism
2. irregular astigmatism
3. prior or ongoing corneal disease or scarring
4. history of ocular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Corneal aberration | 3 months

SECONDARY OUTCOMES:
Visual acuity | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States